CLINICAL TRIAL: NCT03528681
Title: A Phase 3 Multicenter, Prospective, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety and Efficacy of ZS (Sodium Zirconium Cyclosilicate), in Patients With Hyperkalemia-HARMONIZE Asia
Brief Title: A Study to Investigate the Safety and Efficacy of ZS in Patients With Hyperkalemia.
Acronym: HARMONIZE Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9480C00001
Record Dates: First submitted 2018-04-16; First posted 2018-05-18 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium Zirconium Cyclosilicate 10g (Experimental): Suspension administered 10g orally once daily for 28 days after the open label initial phase.
  Interventions: Drug: Sodium Zirconium Cyclosilicate 10g
- Sodium Zirconium Cyclosilicate 5g (Experimental): Suspension administered 5g orally once daily for 28 days after the open label initial phase.
  Interventions: Drug: Sodium Zirconium Cyclosilicate 5g
- Matching Placebo (Placebo Comparator): Suspension administered orally placebo once daily for 28 days after the open label initial phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate 5g — Suspension administered Sodium Zirconium Cyclosilicate 5g orally once daily for 28 days after the open label initial phase with suspension administered Sodium Zirconium Cyclosilicate 10g orally three times per day for at most 2 days.
  Arms: Sodium Zirconium Cyclosilicate 5g
Drug: Sodium Zirconium Cyclosilicate 10g — Suspension administered Sodium Zirconium Cyclosilicate 10g orally once daily for 28 days after the open label initial phase with suspension administered Sodium Zirconium Cyclosilicate 10g orally three times per day for at most 2 days.
  Arms: Sodium Zirconium Cyclosilicate 10g
Drug: Placebo — Suspension administered orally placebo once daily for 28 days after the open label initial phase with suspension administered Sodium Zirconium Cyclosilicate 10g orally three times per day for at most 2 days.
  Arms: Matching Placebo

SUMMARY:
To evaluate the efficacy of two different doses (5 and 10 g) of ZS orally administered once daily (qd) vs placebo in maintaining normokalemia in initially hyperkalemic patients having achieved normokalemia following 24 or 48 hours of initial ZS therapy (10g TID).

DETAILED DESCRIPTION:
This study will be conducted in approximately 35 centers in China. Before patients are randomized to the double-blind phase, they will receive open-label ZS for 24 or 48 hours during the initial phase. It is expected that approximately 490 patients will need to be enrolled, to have approximately 280 patients entered into the open-label initial phase resulting in 250 patients being randomized in the 28-day treatment study phase. Enrolment will be stopped when 250 patients have been initiated with the 28-day randomized treatment study phase.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent (pre-screening consent) prior to any study specific procedures
2. Female and male patients aged ≥18 and ≤ 90 years
3. Provision of informed consent prior to any study specific procedures
4. Two consecutive i-STAT potassium values, measured 60 minutes (± 10 minutes) apart, both ≥ 5.1 mmol/L and measured within 1 day of the first ZS dose on open-label initial phase Day 1
5. Ability to have repeated blood draws or effective venous catheterization
6. Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception for the duration of the study (from the time they sign consent) and for 3 months after the last dose of ZS/matching placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study
2. Participation in another clinical study with an investigational product during the last 3 months
3. Presence of any condition which, in the opinion of the investigator, places the patient at undue risk or potentially jeopardizes the quality of the data to be generated
4. Pseudohyperkalemia signs and symptoms, such as hemolyzed blood specimen due to excessive fist clenching to make veins prominent, difficult or traumatic venepuncture, or history of severe leukocytosis or thrombocytosis
5. Patients treated with lactulose, xifaxan (rifaximin) or other non-absorbed antibiotics for hyperammonemia within 7 days prior to the first dose of study drug
6. Patients treated with resins,calcium acetate,calcium carbonate, or lanthanum carbonate,within 7 days prior to the first dose of study drug
7. Patients with a life expectancy of less than 3 months
8. Patients who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol
9. Female patients who are pregnant, lactating, or planning to become pregnant
10. Patients with diabetic ketoacidosis
11. Known hypersensitivity or previous anaphylaxis to ZS or to components thereof
12. Patients with cardiac arrhythmias that require immediate treatment
13. History of QT prolongation associated with other medications that required discontinuation of that medication.
14. Congenital long QT syndrome
15. Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted
16. QTc(f) > 550 msec
17. Patients on dialysis
18. Patients who are blood donors should not donate blood during the study and for 3 months following their last dose of ZS
19. Patients who need hospitalization after taking blood samples on day 1 of the open-label initial phase

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- China (36):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Dongguan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jilin
  - Research Site, Jinan
  - Research Site, Jingzhou
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xining
  - Research Site, Yangzhou
  - Research Site, Yichang
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zhuzhou
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Chandigarh
  - Research Site, Chennai
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Vijayawada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Liang X, Lu W, Yu X, Cheng H, He Q, Peng Q, Ni Z, Long G, Wang L, Chen W, Li R, Zhao J, Zhang Y, Lisovskaja V, Tang Z. HARMONIZE Asia: A Phase III Randomized Study to Investigate the Efficacy and Safety of Sodium Zirconium Cyclosilicate in Patients with Hyperkalemia in China. Clin Ther. 2024 Sep;46(9):702-710. doi: 10.1016/j.clinthera.2024.07.004. Epub 2024 Aug 6. PMID 39112102
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00001&attachmentIdentifier=a47248d4-96f9-4b78-b851-24164ffe2f86&fileName=D9480C00001_CSP_Redacted.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00001&attachmentIdentifier=6c844f0b-5f48-44bd-9c27-e4539f412cd3&fileName=D9480C00001_SAP_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00001&attachmentIdentifier=bfc960c6-5f05-4753-8c1e-c6bc683bacd6&fileName=D9480C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 35 sites in China.
Pre-assignment Details: The study consisted of two phases, an Open-label initial phase (OLP) and a Randomized treatment phase (RTP).
  270 participants entered OLP, out of these 250 entered RTP & received Placebo, SZC 5g QD, or SZC 10g QD in a 1:2:2 ratio.
Groups:
- Sodium Zirconium Cyclosilicate (SZC) 10g TID: Suspension administered 10g orally 3 times per day for the open-label initial phase
- Sodium Zirconium Cyclosilicate (SZC) 5g QD: Suspension administered 5g orally once daily for 28 days after the open-label initial phase
- Sodium Zirconium Cyclosilicate (SZC) 10g QD: Suspension administered 10g orally once daily for 28 days after the open-label initial phase
- Placebo: Suspension administered placebo orally once daily for 28 days after the open-label initial phase.
Period: Open-Label Phase
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Started | 270 | 0 | 0 | 0
Completed | 256 | 0 | 0 | 0
Not Completed | 14 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0 | 0
Not completed — (Not collected) | 4 | 0 | 0 | 0
Period: Randomized Treatment Phase
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Started | 0 (No subjects were randomized to 10g TID group in the Randomized Treatment Phase) | 100 (100 subjects were randomized to 5g QD group in the Randomized Treatment Phase) | 100 (100 subjects were randomized to 10g QD group in the Randomized Treatment Phase) | 50 (50 subjects were randomized to Placebo group in the Randomized Treatment Phase)
Completed | 0 | 81 | 85 | 38
Not Completed | 0 | 19 | 15 | 12
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 5 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 7 | 4 | 1
Not completed — (Study specific withdrawal criteria) | 0 | 3 | 3 | 4
Not completed — (Not collected) | 0 | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Population: The study consisted of two phases, an Open-label initial phase (OLP) and a Randomized treatment phase (RTP). 270 participants entered OLP, out of these 250 entered RTP & received Placebo, SZC 5g QD or SZC 10g QD in a 1:2:2 ratio.
Groups:
- Sodium Zirconium Cyclosilicate (SZC): Suspension administered 10g orally 3 times per day for the open-label initial phase
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo | Total
Number analyzed (Participants) | 270 | 100 | 100 | 50 | 520
Age, Continuous [Mean (Standard Deviation); unit: Years] — 270 patients entered OLP, out of these 250 entered RTP Population: Two phases reported as separate rows to avoid double counting
  Years
    Randomized treatment phase (RTP): number analyzed (Participants) | 0 | 100 | 100 | 50 | 250
    Randomized treatment phase (RTP) |  | 54.3 (13.92) | 55.6 (14.47) | 59.7 (14.2) | 55.9 (14.28)
    Open-label initial phase (OLP): number analyzed (Participants) | 270 | 0 | 0 | 0 | 270
    Open-label initial phase (OLP) | 56.4 (14.17) |  |  |  | 56.4 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants] — 270 patients entered OLP, out of these 250 entered RTP Population: Two phases reported as separate rows to avoid double counting
  Participants
    Randomized treatment phase (RTP): number analyzed (Participants) | 0 | 100 | 100 | 50 | 250
    Randomized treatment phase (RTP): Female |  | 35 | 40 | 19 | 94
    Randomized treatment phase (RTP): Male |  | 65 | 60 | 31 | 156
    Open-label initial phase (OLP): number analyzed (Participants) | 270 | 0 | 0 | 0 | 270
    Open-label initial phase (OLP): Female | 103 |  |  |  | 103
    Open-label initial phase (OLP): Male | 167 |  |  |  | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — 270 patients entered OLP, out of these 250 entered RTP Population: Two phases reported as separate rows to avoid double counting
  Participants
    Not Hispanic or Latino Randomized treatment phase (RTP): number analyzed (Participants) | 0 | 100 | 100 | 50 | 250
    Not Hispanic or Latino Randomized treatment phase (RTP) |  | 100 | 100 | 50 | 250
    Not Hispanic or Latino Open-label initial phase (OLP): number analyzed (Participants) | 270 | 0 | 0 | 0 | 270
    Not Hispanic or Latino Open-label initial phase (OLP) | 270 |  |  |  | 270

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean S-K Level on Days 8-29
Description: Comparison between placebo and each SZC treatment group (high to low) with regard to the mean S-K level during the randomized treatment phase days 8-29. Mixed-effects models were used to estimate least-squares means.
Time Frame: Days 8 to 29 (Randomized treatment study phase) used for model-based least squares mean computation
Population: Full analysis set - Randomized Treatment Phase
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
mmol/L |  | 4.859 [4.709 to 5.014] | 4.440 [4.304 to 4.580] | 5.225 [5.055 to 5.400]
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; Results are derived from a longitudinal model applied to log-transformed S-K measurements adjusted for treatment, visit, treatment-by-visit interaction and baseline covariates. The back-transformation is to the original scale of the S-K measurement; Test type: Other; p < 0.001, Mixed Models Analysis; Back-transformed mean difference = 0.930, 95% CI 2-sided [0.902 to 0.959]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; Back-transformed mean difference = 0.850, 95% CI 2-sided [0.825 to 0.876]

2. Secondary Outcome: Percentage of Patients Who Achieve Normokalemia
Description: Percentage of patients who achieve normokalemia during the open label initial phase at 24 hours and at the end of the open label phase. End of OLP is defined as Day 2 (24 hours post first dose) or Day 3 (48 hours post first dose) depending on when the subject achieved normokalemia based on the pre-dose i-STAT potassium level. The results in the table below are presented for OLP.
Time Frame: Through open label initial phase
Population: Full analysis set - Open Label Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 261 | 0 | 0 | 0
Participants
  Normokalemic at 24h | 180 |  |  |
  Normokalemic at End of OLP | 228 |  |  |

3. Secondary Outcome: Exponential Rate of Change in S-K Levels
Description: Exponential rate of change in S-K levels (blood) during the open-label initial phase 24 hours post-dose. Least Square Mean corresponds to the exponential rate of change i.e. the slope (for time) in terms of log-transformed S-K levels. The results in the table below are presented for OLP.
Time Frame: Through 24 hours post-dose in the initial phase
Population: Full analysis set - Open Label Phase
Measure: Least Squares Mean (Standard Error); unit: log(mmol/L)/h
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 270 | 0 | 0 | 0
log(mmol/L)/h | -0.0051 (0.00027) |  |  |

4. Secondary Outcome: Absolute Change From Baseline in S-K Levels
Description: Absolute change from baseline in S-K levels at all measured time intervals. End of OLP is defined as Day 2 (24 hours post first dose) or Day 3 (48 hours post first dose) depending on when the subject achieved normokalemia based on the pre-dose i-STAT potassium level. The results in the table below are presented for OLP.
Time Frame: Through open label initial phase
Population: Full analysis set - Open Label Phase
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 261 | 0 | 0 | 0
mmol/L
  OLP - 24 hours | -0.936 (0.377) |  |  |
  End of OLP | -1.107 (0.466) |  |  |

5. Secondary Outcome: Percentage Change From Baseline in S-K Levels
Description: Percentage change from baseline in S-K levels at all measured time intervals. End of OLP is defined as Day 2 (24 hours post first dose) or Day 3 (48 hours post first dose) depending on when the subject achieved normokalemia based on the pre-dose i-STAT potassium level. The results in the table below are presented for OLP.
Time Frame: Through open label initial phase
Population: Full analysis set - Open Label Phase
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 261 | 0 | 0 | 0
Percentage
  OLP - 24 hours | -15.880 (5.980) |  |  |
  End of OLP | -18.588 (6.701) |  |  |

6. Secondary Outcome: Proportion of Patients Who Remain Normokalemic During RTP
Description: Proportion of patients who remain normokalemic (as defined by S-K between 3.5-5.0 mmol/l, inclusive) during RTP (Day 8 to Day 29). The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment study phase day 8-29
Population: Full analysis set - Randomized Treatment Phase
Measure: Number; unit: Average probability
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 99 | 98 | 50
Average probability |  | 0.596 | 0.818 | 0.279
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; Test type: Other — The analysis uses a generalized mixed model which includes a random intercept and logit link. The model includes all S-K data values collected at the scheduled visits between Days 8-29, dichotomized as normal and abnormal, as response variables, and baseline covariates. Placebo is the reference group; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 3.80, 95% CI 2-sided [2.17 to 6.67]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; The analysis uses a generalized mixed model which includes a random intercept and logit link. The model includes all S-K data values collected at the scheduled visits between Days 8-29, dichotomized as normal and abnormal, as response variables, and baseline covariates. Placebo is the reference group; Test type: Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 11.63, 95% CI 2-sided [6.45 to 21.00]

7. Secondary Outcome: Proportion of Normokalemic Patients at the End of RTP
Description: Proportion of normokalemic patients (as defined by S-K between 3.5-5.0 mmol/l, inclusive). The results in the table below are presented for RTP.
Time Frame: The end of 28-day randomized treatment study phase
Population: Full analysis set - Randomized Treatment Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 80 | 85 | 38
Participants |  | 47 | 65 | 14
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; Test type: Other — The model included normokalaemia status (yes, no) on Day 29 as binary response variables, and baseline covariates. Placebo is the reference group; p = 0.035, Regression, Logistic; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.07 to 6.05]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; The model included normokalaemia status (yes, no) on Day 29 as binary response variables, and baseline covariates. Placebo is the reference group; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.25, 95% CI 2-sided [2.56 to 15.27]

8. Secondary Outcome: Days Patients Remain Normokalemic
Description: The number of days patients remain normokalemic during days 8-29 of the randomized treatment study phase. The results in the table below are presented for RTP.
Time Frame: Through days 8-29 of the randomized treatment phase.
Population: Full analysis set - Randomized Treatment Phase
Measure: Least Squares Mean (Standard Error); unit: Day
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 99 | 98 | 50
Day |  | 9.11 (1.413) | 14.54 (1.397) | 3.40 (1.473)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; Results derived from a linear regression model with the following covariates: treatment group; baseline S-K values (Open-label phase and Randomized treatment phase); baseline eGFR; age category; country; baseline RAAS inhibitor, chronic kidney disease, heart failure, and diabetes mellitus statuses; Test type: Other; p < 0.001, Regression, Linear; Median Difference (Final Values) = 5.72, 95% CI 2-sided [3.13 to 8.31]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Other; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 11.14, 95% CI 2-sided [8.57 to 13.71]

9. Secondary Outcome: Mean Change in S-K Levels
Description: The mean change in S-K levels evaluated relative to the RTP baseline. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full analysis set - Randomized Treatment Phase
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 98 | 99 | 50
mmol/L
  Day 2 change from RTP baseline: number analyzed (Participants) | 0 | 84 | 86 | 41
  Day 2 change from RTP baseline |  | -0.04 (0.299) | -0.15 (0.314) | 0.02 (0.315)
  Day 5 change from RTP baseline: number analyzed (Participants) | 0 | 98 | 99 | 49
  Day 5 change from RTP baseline |  | 0.09 (0.434) | -0.27 (0.464) | 0.40 (0.423)
  Day 8 change from RTP baseline: number analyzed (Participants) | 0 | 96 | 98 | 50
  Day 8 change from RTP baseline |  | 0.20 (0.481) | -0.29 (0.541) | 0.53 (0.485)
  Day 12 change from RTP baseline: number analyzed (Participants) | 0 | 89 | 96 | 45
  Day 12 change from RTP baseline |  | 0.25 (0.539) | -0.23 (0.597) | 0.67 (0.452)
  Day 15 change from RTP baseline: number analyzed (Participants) | 0 | 91 | 93 | 48
  Day 15 change from RTP baseline |  | 0.26 (0.557) | -0.24 (0.581) | 0.67 (0.494)
  Day 19 change from RTP baseline: number analyzed (Participants) | 0 | 84 | 88 | 41
  Day 19 change from RTP baseline |  | 0.41 (0.606) | -0.19 (0.616) | 0.61 (0.506)
  Day 22 change from RTP baseline: number analyzed (Participants) | 0 | 85 | 87 | 43
  Day 22 change from RTP baseline |  | 0.32 (0.543) | -0.13 (0.538) | 0.62 (0.536)
  Day 26 change from RTP baseline: number analyzed (Participants) | 0 | 76 | 81 | 41
  Day 26 change from RTP baseline |  | 0.22 (0.556) | -0.05 (0.627) | 0.55 (0.447)
  Day 29 change from RTP baseline: number analyzed (Participants) | 0 | 80 | 85 | 38
  Day 29 change from RTP baseline |  | 0.23 (0.494) | 0.01 (0.578) | 0.47 (0.520)
  EOS change from RTP baseline: number analyzed (Participants) | 0 | 78 | 82 | 36
  EOS change from RTP baseline |  | 0.57 (0.499) | 0.67 (0.688) | 0.55 (0.667)

10. Secondary Outcome: Mean Percent Change in S-K Levels
Description: The mean percent change in S-K levels evaluated relative to the RTP baseline. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full analysis set - Randomized Treatment Phase
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 98 | 99 | 50
Percent change
  Day 2 change from RTP baseline: number analyzed (Participants) | 0 | 84 | 86 | 41
  Day 2 change from RTP baseline |  | -0.81 (6.308) | -3.13 (6.627) | 0.41 (6.670)
  Day 5 change from RTP baseline: number analyzed (Participants) | 0 | 98 | 99 | 49
  Day 5 change from RTP baseline |  | 2.10 (9.009) | -5.57 (9.688) | 8.56 (8.989)
  Day 8 change from RTP baseline: number analyzed (Participants) | 0 | 96 | 98 | 50
  Day 8 change from RTP baseline |  | 4.45 (10.260) | -6.05 (11.352) | 11.24 (9.989)
  Day 12 change from RTP baseline: number analyzed (Participants) | 0 | 89 | 96 | 45
  Day 12 change from RTP baseline |  | 5.55 (11.564) | -4.65 (12.604) | 14.39 (9.908)
  Day 15 change from RTP baseline: number analyzed (Participants) | 0 | 91 | 93 | 48
  Day 15 change from RTP baseline |  | 5.85 (11.840) | -4.85 (12.107) | 14.50 (10.775)
  Day 19 change from RTP baseline: number analyzed (Participants) | 0 | 84 | 88 | 41
  Day 19 change from RTP baseline |  | 9.01 (13.285) | -3.76 (12.797) | 13.34 (11.266)
  Day 22 change from RTP baseline: number analyzed (Participants) | 0 | 85 | 87 | 43
  Day 22 change from RTP baseline |  | 7.09 (11.952) | -2.59 (11.292) | 13.15 (11.686)
  Day 26 change from RTP baseline: number analyzed (Participants) | 0 | 76 | 81 | 41
  Day 26 change from RTP baseline |  | 5.12 (12.130) | -0.76 (13.278) | 11.95 (9.809)
  Day 29 change from RTP baseline: number analyzed (Participants) | 0 | 80 | 85 | 38
  Day 29 change from RTP baseline |  | 5.24 (10.941) | 0.48 (12.142) | 10.20 (11.438)
  EOS change from RTP baseline: number analyzed (Participants) | 0 | 78 | 82 | 36
  EOS change from RTP baseline |  | 12.42 (11.054) | 14.47 (14.797) | 11.74 (14.477)

11. Secondary Outcome: Least Square Mean Changes in S-Aldo and P-Renin Levels
Description: Comparison between placebo and each SZC treatment group (high to low) with regard to the mean S-Aldo and P-Renin levels during the randomized treatment phase days 15-29.
Time Frame: Through 28 day randomized treatment study phase day 15-29
Population: Full analysis set - Randomized Treatment Phase
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 88 | 92 | 46
pmol/L
  S-Aldo |  | -21.926 [-80.492 to 36.640] | -53.945 [-112.189 to 4.300] | 83.322 [22.519 to 144.124]
  P-Renin: number analyzed (Participants) | 0 | 86 | 90 | 44
  P-Renin |  | -0.348 [-0.484 to -0.212] | -0.424 [-0.559 to -0.288] | -0.362 [-0.505 to -0.218]
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; S-Aldo Results derived from a longitudinal mixed model adjusted for treatment, visit, treatment-by-visit interaction and baseline covariates; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -105.248, 95% CI 2-sided [-161.293 to -49.203]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -137.267, 95% CI 2-sided [-192.596 to -81.937]
Statistical Analysis 3: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; P-Renin Results derived from a longitudinal mixed model adjusted for treatment, visit, treatment-by-visit interaction and baseline covariates; Test type: Other; p = 0.839, Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.120 to 0.147]
Statistical Analysis 4: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Other; p = 0.355, Mixed Models Analysis; Mean Difference (Final Values) = -0.062, 95% CI 2-sided [-0.195 to 0.070]

12. Secondary Outcome: Hyperkalaemia at Day 29
Description: The number of patients with hyperkalaemia at day 29. The results in the table below are presented for RTP.
Time Frame: Day 29
Population: Full analysis set - Randomized Treatment Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 100 | 99 | 50
Participants |  | 77 | 50 | 48

13. Secondary Outcome: Percentage of Patients Without Hyperkalemia
Description: Kaplan-Meier estimate at Day 29 of percentage of patients without hyperkalemia. The results in the table below are presented for RTP.
Time Frame: Day 29 of randomized treatment phase
Population: Full analysis set - Randomized Treatment Phase
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
Number analyzed (Participants) | 0 | 100 | 99 | 50
Percentage |  | 20.3 [12.8 to 29.0] | 47.1 [36.5 to 57.0] | 4.0 [0.7 to 12.1]
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) 5g QD vs Placebo; The model included time to reoccurrence of hyperkalaemia as response variable (event: hyperkalaemia or discontinue treatment in RTP due to high S-K levels), baseline eGFR, OLP and RTP baseline S-K values as well as age (< 55, 55-64, > 64 years) and baseline binary indicators for RAASi, chronic kidney disease, heart failure, and diabetes mellitus as covariates. Placebo is the reference group; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.27 to 0.57]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (SZC) 10g QD vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.10 to 0.25]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the main study informed consent (Day 1, Visit 3) throughout the treatment period and including the End of Study (EOS) visit. Serious Adverse Events were collected from the time of the optional Pre-screening informed consent (Visit 1) throughout the treatment period and including the EOS visit. Maximum duration of treatment was 8 days for open-label initial phase and 30 days for the randomized treatment phase.
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g TID | Sodium Zirconium Cyclosilicate (SZC) 5g QD | Sodium Zirconium Cyclosilicate (SZC) 10g QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/100 | 0/100 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/270 | 6/100 | 3/100 | 1/50
Other Adverse Events (participants affected / at risk) | 38/270 | 48/100 | 42/100 | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) 10g TID (N=270) | Sodium Zirconium Cyclosilicate (SZC) 5g QD (N=100) | Sodium Zirconium Cyclosilicate (SZC) 10g QD (N=100) | Placebo (N=50)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) 10g TID (N=270) | Sodium Zirconium Cyclosilicate (SZC) 5g QD (N=100) | Sodium Zirconium Cyclosilicate (SZC) 10g QD (N=100) | Placebo (N=50)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Secondary hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Orbital swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (7) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (5) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 8 (8) | 12 (13) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (5) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram p wave biphasic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram q wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram st-t segment abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (5) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT03528681/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03528681/SAP_001.pdf